CLINICAL TRIAL: NCT06144723
Title: Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetic and the Therapeutic Potential of HS-20105 for Injection in Patients With Advanced Solid Tumors.
Brief Title: Study of HS-20105 for Injection in Patients With Advanced Solid Tumors.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20105-101
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; HS-20105; Trop-2; ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20105 Phase Ia (Dose escalation) (Experimental): Patients with advanced solid tumors will be enrolled and receive HS-20105 of various dose strengths until the end of the study in the absence of unacceptable toxicities and disease progression.
  Interventions: Drug: HS-20105
- HS-20105 Phase Ib (Dose expansion) (Experimental): Depending on data obtained from the dose escalation, dose expansion may proceed with multiple cohorts in subjects with advanced solid tumors. Patients enrolled will receive HS-20105 until the end of the study in the absence of unacceptable toxicities and disease progression. The recommended doses from the dose escalation will be further explored.
  Interventions: Drug: HS-20105

INTERVENTIONS:
Drug: HS-20105 — Administered intravenously every 21 days.

SUMMARY:
HS-20105 is a novel antibody-drug conjugate (ADC) targeting Trop-2. This first-in-human trial is aimed to assess the maximum tolerated dose (MTD) and dose limiting toxicity (DLT), to evaluate the pharmacokinetics (PK), safety and preliminary anti-tumor activity of HS-20105 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase I clinical study evaluating the safety, tolerability, PK, and efficacy of HS-20105 in patients with advanced solid tumors. The study includes Phase Ia (dose escalation) and Phase Ib (dose extension). Phase Ia will conduct a dose escalation using the "Rolling 6" design in advanced solid tumor patients who have failed or are unable to tolerate standard treatment, to evaluate the safety, tolerability, PK characteristics, and efficacy of HS-20105. The subsequent Phase Ib study will be conducted in certain population to evaluate the preliminary efficacy of HS-20105 at different doses and in different populations.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged more than or equal to (≥) 18 years.
* Advanced solid tumor patients confirmed by histology or cytology for who that standard treatment is failed or intolerable.
* Patients have at least one target lesion according to RECEST 1.1. The requirements for target lesions are: measurable lesions without local treatment such as irradiation, or with definite progress after local treatment, with the longest diameter ≥ 10 mm in the baseline period (in case of lymph nodes, the shortest axis ≥ 15 mm is required). Patients with only brain and/or bone lesions as target lesions will not be included.
* Fresh or archived tumor tissue samples need to be provided (fresh samples are preferred, and tumor tissue samples within 2 years before the first administration can be accepted; the sample type is formalin fixed, paraffin embedded [FFPE] tumor tissue block or FFPE slides).
* ECOG performance status was 0-1 and did not deteriorate in the previous 2 weeks.
* Estimated life expectancy greater than (>) 12 weeks.
* Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 6 months after the last dose. Likewise, men also consent to use adequate contraceptive method within the same time limit.
* Females must have the evidence of non-childbearing potential.
* Sign informed consent form.

Exclusion Criteria:

* Has received or is currently undergoing the following treatment:

  1. Previously or current treatment with drugs targeting Trop-2 or other ADC drugs conjugated with HS-9265;
  2. Received traditional Chinese medicine therapy with anti-tumor indications within 2 weeks prior to the first administration of HS-20105;
  3. Received cytotoxic chemotherapy drugs or other anti-tumor system therapies (including endocrine therapy, molecular targeted therapy, or biological therapy) within 3 weeks prior to the first administration of HS-20105;
  4. Received macromolecular anti-tumor drugs or experimental drug therapy within 4 weeks before the first administration of HS-20105;
  5. Received local radiotherapy within 2 weeks before the first administration of HS-20105; Received more than 30% of bone marrow irradiation or extensive radiation therapy within 4 weeks before the first administration of HS-20105;
  6. Received major surgery within 4 weeks before the first administration of HS-20105.
  7. Received strong inhibitors or inducers of CYP3A4, CYP2D6, P-gp or BCRP, or drugs with narrow treatment windows for CYP3A4, CYP2D6, P-gp or BCRP sensitive substrates, have been used.
  8. Receiving medication that is known to prolong the QT interval or may lead to torsade de pointes.
* Existing abnormal CTCAE ≥ grade 2 resulted from previous treatment.
* History of other malignancy.
* Uncontrolled pleural, ascites or pericardial effusion.
* Known and unstable central nervous system metastases.
* Inadequate bone marrow reserve or serious organ dysfunction.
* Severe, uncontrolled, or active cardiovascular disease.
* Severe or poorly controlled diabetes.
* Severe or poorly controlled hypertension.
* Clinically significant bleeding symptoms within 1 month before the first administration of HS-20105.
* Serious thrombosis events within 3 months before the first administration of HS-20105.
* Serious infection within 4 weeks before the first administration of HS-20105.
* Received continuous glucocorticoid treatment for more than 7 days within 28 days before the first administration of HS-20105.
* Active infectious disease.
* Hepatic encephalopathy, hepatorenal syndrome, or ≥ Child-Pugh B-grade cirrhosis.
* Serious or uncontrolled eye disease.
* Moderate to severe lung diseases that may interfere with the detection or management of drug-related pulmonary toxicity and seriously affect respiratory function.
* Severe neurological or mental disorders that can interfere with assessment.
* Pregnant women, breastfeeding women or woman who has a child-bearing plan during the study.
* History of hypersensitivity to any active or inactive ingredient of HS-20105.
* The subject who is unlikely to comply with study procedures, restrictions, or requirements, judged by the investigator
* The subject whose safety cannot be ensured or study assessments would be interfered, judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: MTD or maximum applicable dose (MAD) of HS-20105 | Up to12 months.
  Number of participants with DLT.
Phase Ib: Efficacy of HS-20105 | Up to 24 months.
  Objective response rate (ORR) according to response evaluation criteria in solid tumors (RECIST) 1.1 by investigator's assessment.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | Up to 36 months.
  Incidence of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Disease control rate (DCR) | Up to 24 months.
  The percentage of patients who have achieved complete response, partial response, and stable disease, according to response evaluation criteria in solid tumors (RECIST) 1.1 by investigator's assessment.
Duration of response (DoR) | Up to 24 months.
  The time from complete or partial response to disease progression or death, according to response evaluation criteria in solid tumors (RECIST) 1.1 by investigator's assessment.
Progression-free survival (PFS) | Up to 24 months.
  Progression free survival is defined as the duration of time from study entry to time of progression, death, or is censored at date of last disease assessment.
Overall survival (OS) | Up to 3 years
  Overall survival is defined as the duration of time from study entry to death or the date of last contact.
Maximum plasma concentration (Cmax) | Up to 24 months.
  Cmax is defined as maximum observed serum concentration obtained directly from the observed concentration-time data.
Time of maximum concentration (Tmax) | Up to 24 months.
  Tmax is defined as the time required for a drug to reach peak concentration in plasma.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) | Up to 24 months.
  Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration.
Elimination half-life (T1/2) | Up to 24 months.
  T1/2 is defined as apparent terminal elimination half-life (h).
Anti-drug antibodies (ADA) of HS-20105 | Up to 24 months.
  Number of participants who are positive for ADA will be reported..